CLINICAL TRIAL: NCT06464419
Title: Ultrasonographic Evaluation of Optic Nerve Sheath Diameter in Patients Undergoing Retrograde Intrarenal Surgery in the Lithotomy Position
Brief Title: Effect of Lithotomy Position on Optic Nerve Sheath Diameter
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14408
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-06

CONDITIONS: Optic Nerve Cup; Intracranial Pressure Increase
Keywords: ultrasonography, lithotomy position
MeSH Terms: conditions — Intracranial Hypertension | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who will undergo RIRS surgery: Patients who will undergo RIRS surgery in the lithotomy position
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — Measurement of optic nerve sheath diameter by ultrasound

SUMMARY:
In this study, the effect of increased venous return and increased intra-abdominal pressure on intracranial pressure in the lithotomy position was evaluated.

DETAILED DESCRIPTION:
In the lithotomy position, it is possible that venous return in the lower extremities increases and intra-abdominal pressure increases due to the position. At the same time, it is possible that the intracompartmental pressure in the extremities increases because the venous structure is compressed by placing the lower extremities on supports. Considering both conditions, it is predicted that there may be an increase in the optic nerve sheath diameter due to increased intracranial pressure in patients placed in the lithotomy position. The aim of this study is to investigate the effect of the position on intracranial pressure by ultrasonographically evaluating the optic nerve sheath diameter in the lithotomy position.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give informed consent
* Patients who will undergo retrograde intrarenal surgery
* Patients who are fully oriented and cooperative
* ASA I-II patients
* Patients between the ages of 18-65

Exclusion Criteria:

* Disoriented and uncooperative patients
* Patients with BMI>30
* Patients who have had previous intracranial surgery
* Patients who have had eye surgery before
* Patients allergic to the pharmacological agents used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 52 patients, ASA I-II, aged between 18-65, who are scheduled for elective RIRS surgery under general anesthesia will be included.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Effect of lithotomy position on optic nerve sheath diameter | intraoperative and postoperative 10 minutes
  In patients in the lithotomy position, the linear probe of the ultrasound will be placed on the patient's upper eyelid in a transverse and longitudinal manner without applying compression, and the optic nerve's entry into the orbit will be visualized and measured. The increase in the optic nerve sheath diameter will be recorded by measuring at 7 different times in total.Before general anesthesia (t1), 3 minutes (min.) (t2) and 5 min. (t3) after general anesthesia, 3 min. (t4) and 5 min. (t5) after lithotomy position was given, before lithotomy position was corrected (t6) and when 10 minutes after patients go to the recovery room (t7).

CONTACTS AND LOCATIONS:
Overall Officials: Cansu Ekici, Study Director — EtlikCityHospital
Locations (1):
- EtlikCityHospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Result] Maissan IM, Dirven PJ, Haitsma IK, Hoeks SE, Gommers D, Stolker RJ. Ultrasonographic measured optic nerve sheath diameter as an accurate and quick monitor for changes in intracranial pressure. J Neurosurg. 2015 Sep;123(3):743-7. doi: 10.3171/2014.10.JNS141197. Epub 2015 May 8. PMID 25955869
- [Result] Besir A, Tugcugil E. Effects of tourniquet usage in lower extremity surgery on optic nerve sheath diameter. Turk J Med Sci. 2018 Oct 31;48(5):980-984. doi: 10.3906/sag-1803-132. PMID 30384564
- [Result] Blecha S, Harth M, Schlachetzki F, Zeman F, Blecha C, Flora P, Burger M, Denzinger S, Graf BM, Helbig H, Pawlik MT. Changes in intraocular pressure and optic nerve sheath diameter in patients undergoing robotic-assisted laparoscopic prostatectomy in steep 45 degrees Trendelenburg position. BMC Anesthesiol. 2017 Mar 11;17(1):40. doi: 10.1186/s12871-017-0333-3. PMID 28284189